CLINICAL TRIAL: NCT03746314
Title: Supportive Care Service Availability for Cancer Caregivers in Community Oncology Practices
Acronym: Caregivers
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00054509; WF-1803CD (Other: NCI); 3UG1CA189824-04S1 (NIH); NCI-2018-02596 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2018-11-16; First posted 2018-11-19 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Supportive Care
Keywords: Caregivers; Oncology; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Supportive Care Leader: A staff member who is knowledgeable about supportive care services for adult oncology patients.
- Oncology Providers: Physicians, nurses, physicians assistants, nurse practitioners who routinely provide cancer care to adult oncology patients.

SUMMARY:
The purpose of this study is to understand current practices for engaging with informal (unpaid) caregivers of patients with cancer, characterize the availability of supportive care services, and assess the perspectives of multi-disciplinary oncology health care providers regarding identifying and supporting caregivers.

DETAILED DESCRIPTION:
The primary goals of this study are to: 1) estimate the prevalence of: a) caregiver identification practices, b) psychosocial and/or needs assessment practices for caregivers, and c) the availability of and funding models for supportive care services for caregivers at community oncology practices (Objective 1), and 2) assess the perspectives of multi-disciplinary oncology health care providers regarding: a) perceived responsibility for, and barriers to, assessing and supporting caregivers, b) the importance of and self-efficacy in communicating with caregivers, and c) preferences regarding systems approaches to assess and meet caregivers' needs (Objective 2). Additionally, we will explore various practice and provider -level factors that are associated with the listed outcomes in objectives 1 and 2 respectively (Objective 3a and 3b). This study is estimated to enroll 138 Supportive Care Leaders (e.g., Director of Psychosocial Oncology, Supportive Care Services, or Cancer Patient Support) and 690 multidisciplinary Oncology Providers including physicians, nurses, and physician assistants/nurse practitioners. Participants will complete a one-time web-based survey (estimated at 15-20 minutes to complete). The supportive care leader survey will capture: (1) practice characteristics including caregiver identification and psychosocial assessment practices and preferences; supportive care resources; practice structure; practice technology resources; and status of the Caregiver Advise Record and Enable (CARE) Act. The oncology provider survey will capture: (1) provider skills in caregiver communication; perceived responsibility, knowledge and skills, and awareness of resources for meeting caregiver needs; barriers to meeting caregiver needs; provider characteristics; and system intervention preferences.

For data capture regarding supportive care leaders (Objective 1 and 3a), this will be a convenience sample of responders from all WF NCORP sites, therefore no randomization or stratification is necessary.

Regarding objectives pertaining to oncology providers (Objective 2 and 3b), participating sites with corresponding supportive care leaders will identify an appropriate supportive care leader to generate 3 lists of providers: 1) physicians, 2) nurses, and 3) physician assistants/nurse practitioners who routinely provide cancer care (Oncology Care Provider Identification Form, Appendix B). Using previous Landscape data regarding oncology physicians, we estimate that 50% of practice groups have 1-9 oncology physicians, 25% have 10-20, and 25% have 20+ physicians. After practices respond with lists of physicians, nurses, and physician assistants/nurse practitioners, we will classify each site as small, medium, and large using the criteria for physicians listed above. Assuming similar distributions as seen in Landscape, we will randomly sample 4, 12, and 20 total providers at small, medium, and large sites respectively. With approximately 50% of practices participating, we plan to target a weighted average of 10 providers per practice with the goal of a weighted average of 5 completed provider surveys (50% response/practice) for a total of 690 providers included in objective 2 (sample size justification follows in section 9.3). In addition, we will stratify and proportionally allocate by provider types identified at each site using self-weighting samples supplied in their lists of providers. Therefore of those randomly sampled, we will target roughly the same proportion of physicians, nurses, and PA/nurse practitioners as identified from their site administrator. Coordinators at each NCORP practice will provide e-mail addresses only for randomly selected providers (selected numbers from a numbered list), based on the size of the center and stratified proportional to provider types.

ELIGIBILITY:
Inclusion Criteria:

* NCI Community Oncology Research Program (NCORP) components/subcomponents providing care to adult oncology patients.
* NCORP components/subcomponents willing to: a) identify a supportive care leader knowledgeable about supportive care services that may be available to the practice and b) assist with the identification and recruitment of oncology providers for a brief provider survey.
* NCORP components/subcomponents who share staff and supportive care services may participate as a single practice group
* A staff member at each site who is most knowledgeable about supportive care services for adult oncology patients (e.g., Director of Manger of Psychosocial Oncology, Supportive Care Services, or Cancer Patient Support). If an administrator or leader cannot be identified, the nurse manager or clinic director will be asked to identify a staff member most knowledgeable about psychosocial or supportive care services for adult oncology patients or complete the survey himself or herself.
* Must be a physician, nurse, or physician assistant/nurse practitioner, who routinely provides cancer care to adult oncology patients, including medical, radiation and surgical oncologists or physician assistants (PAs), nurse practitioners (NPs), and nurses who work in oncology settings.
* Must have been in practice at component/subcomponent for at least 6 months.

Exclusion Criteria:

* Component/subcomponent exclusively care for pediatric oncology patients. Given the distinct caregiver experience and needs of caregivers of pediatric oncology patients, we are not including components/sub-components that exclusively provide care for pediatric oncology patients.
* Providers in practice less than 6 months.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be open to all Adult NCORP Components and Sub-components. Participants will include supportive care leaders (staff member who is most knowledgeable about supportive care services) and multidisciplinary oncology providers (physicians, nurses, and physician assistants/nurse practitioners who routinely provide cancer care and have been in practice at component/subcomponent for at least 6 months).
Sampling Method: Probability Sample
Enrollment: 910 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Percent of Practices that have Mechanisms in Place to Identify Primary Caregivers | Included in One-Time Web-Based Survey; Up to 20 minutes Total
  Practices that have a mechanism in place to identify and document a primary, informal caregiver for cancer patients will be identified by using the following Landscape 2017 Survey item: "Does your practice have a mechanism in place to identify and document a primary, informal (unpaid) caregiver for cancer patients?"
Percent of Practices that have Mechanisms in Place to Provide Psychosocial and/or Needs Assessments for Caregivers | Included in One-Time Web-Based Survey; Up to 20 minutes Total
  Methods, documentation, settings and timing will be collected and assessed from practices that have mechanisms in place to identify primary caregivers.
Percent of Practices that have Availability of and Funding Models for Supportive Care Services | Included in One-Time Web-Based Survey; Up to 20 minutes Total
  Percent of practices that have availability of and funding models for supportive care services provided to patients only, caregivers only, or both patients and caregivers will be assessed using items and content adapted from the Service Availability Measure and the Supportive Care Resources surveys.
Providers' Perceived Responsibility per SPARCCS | Included in One-Time Web-Based Survey; Up to 20 minutes Total
  Questions used to collect perceived responsibility are adapted from the Survey of Physician Attitudes Regarding the Care of Cancer Survivors (SPARCCS) on a scale of 0-4, "strongly disagree" to "strongly agree". These questions assess modifiable constructs that can be targeted for systems level interventions including: 1) questions assessing perceived responsibility for assessing caregivers; 2) questions assessing skills and time to support caregivers; and 3) questions assessing awareness of resources for caregivers in practice and community.
Providers' Perceived Responsibility for Barriers to Meeting Caregiver Needs | Included in One-Time Web-Based Survey; Up to 20 minutes Total
  Barriers to meeting needs of caregivers will be assessed using a 20-item tool designed by our team in prior research which was adapted for this study. Providers will report the extent to which they believe each barrier (e.g., time, lack of specialized staff, reimbursement) impacts service delivery for caregivers on a scale of 0-3, "not a barrier at all" to "Major barrier".
Providers' Ratings of Perceived Importance of Skills in Caregiver Communication | Included in One-Time Web-Based Survey; Up to 20 minutes Total
  Providers' perceived skills in caregiver communication assesses providers' perceived importance, self-efficacy, and need for more training in 4 caregiver communication skills: 1) educating caregivers about ways to support a care recipient during treatment and recovery, 2) detecting when caregivers are anxious, depressed, or overwhelmed, 3) providing information about resources available to support caregivers, 4) assessing problems between caregivers and patients that impact patient treatment or recovery (15 items). These 15 items are adapted from a provider patient communication instrument on a scale of 0-4, "not at all" to "extremely/very much".
Providers' System Intervention Preferences | Included in One-Time Web-Based Survey; Up to 20 minutes Total
  Providers' system intervention preferences will be assessed with 13 items assessing providers' preferences for offering different types of system interventions on a scale of 0-4, "not alt all interested" to "extremely interested"; 12 items assessing willingness and preferences for receiving training in each type of systems intervention on a scale of 0-2, "definitely" to "no".

CONTACTS AND LOCATIONS:
Overall Officials: Chandylen Nightingale, PhD, Principal Investigator — Wake Forest University Health Sciences; Katherine Sterba, PhD, Principal Investigator — Medical University of South Carolina
Locations (272):
- United States (272):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Reid Health, Richmond, Indiana
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Statesville, Statesville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, Wilkesboro, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Memorial Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Bon Secours Health Center at Harbour View, Suffolk, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration.
Access Criteria: upon request to NCORP@wakehealth.edu

REFERENCES:
- [Background] Kent EE, Rowland JH, Northouse L, Litzelman K, Chou WY, Shelburne N, Timura C, O'Mara A, Huss K. Caring for caregivers and patients: Research and clinical priorities for informal cancer caregiving. Cancer. 2016 Jul 1;122(13):1987-95. doi: 10.1002/cncr.29939. Epub 2016 Mar 17. PMID 26991807
- [Background] Northouse LL, Katapodi MC, Schafenacker AM, Weiss D. The impact of caregiving on the psychological well-being of family caregivers and cancer patients. Semin Oncol Nurs. 2012 Nov;28(4):236-45. doi: 10.1016/j.soncn.2012.09.006. PMID 23107181
- [Background] Kim Y, Kashy DA, Spillers RL, Evans TV. Needs assessment of family caregivers of cancer survivors: three cohorts comparison. Psychooncology. 2010 Jun;19(6):573-82. doi: 10.1002/pon.1597. PMID 19582798
- [Background] Northouse L, Williams AL, Given B, McCorkle R. Psychosocial care for family caregivers of patients with cancer. J Clin Oncol. 2012 Apr 10;30(11):1227-34. doi: 10.1200/JCO.2011.39.5798. Epub 2012 Mar 12. PMID 22412124
- [Background] Nightingale CL, Sterba KR, Tooze JA, Milliron BJ, Tetrick LA, Paek MS, Weaver KE. Vulnerable characteristics and interest in wellness programs among head and neck cancer caregivers. Support Care Cancer. 2016 Aug;24(8):3437-45. doi: 10.1007/s00520-016-3160-z. Epub 2016 Mar 19. PMID 26992407
- [Background] Hashemi-Ghasemabadi M, Taleghani F, Yousefy A, Kohan S. Transition to the new role of caregiving for families of patients with breast cancer: a qualitative descriptive exploratory study. Support Care Cancer. 2016 Mar;24(3):1269-76. doi: 10.1007/s00520-015-2906-3. Epub 2015 Aug 26. PMID 26306519
- [Background] Mollica MA, Litzelman K, Rowland JH, Kent EE. The role of medical/nursing skills training in caregiver confidence and burden: A CanCORS study. Cancer. 2017 Nov 15;123(22):4481-4487. doi: 10.1002/cncr.30875. Epub 2017 Jul 20. PMID 28727147
- [Background] Braun M, Mikulincer M, Rydall A, Walsh A, Rodin G. Hidden morbidity in cancer: spouse caregivers. J Clin Oncol. 2007 Oct 20;25(30):4829-34. doi: 10.1200/JCO.2006.10.0909. PMID 17947732
- [Background] Butow PN, Price MA, Bell ML, Webb PM, deFazio A; Australian Ovarian Cancer Study Group; Australian Ovarian Cancer Study Quality Of Life Study Investigators; Friedlander M. Caring for women with ovarian cancer in the last year of life: a longitudinal study of caregiver quality of life, distress and unmet needs. Gynecol Oncol. 2014 Mar;132(3):690-7. doi: 10.1016/j.ygyno.2014.01.002. Epub 2014 Jan 11. PMID 24423880
- [Background] Hammer SL, Clark K, Grant M, Loscalzo MJ. Seventeen years of progress for supportive care services: A resurvey of National Cancer Institute-designated comprehensive cancer centers. Palliat Support Care. 2015 Aug;13(4):917-25. doi: 10.1017/S1478951514000601. Epub 2014 Jul 3. PMID 24992515
- [Background] Ferrell B, Wittenberg E. A review of family caregiving intervention trials in oncology. CA Cancer J Clin. 2017 Jul 8;67(4):318-325. doi: 10.3322/caac.21396. Epub 2017 Mar 20. PMID 28319263
- [Background] Coleman EA. Family caregivers as partners in care transitions: The caregiver advise record and enable act. J Hosp Med. 2016 Dec;11(12):883-885. doi: 10.1002/jhm.2637. Epub 2016 Jul 5. PMID 27378748
- [Background] Whitlatch CJ, Schur D, Noelker LS, Ejaz FK, Looman WJ. The stress process of family caregiving in institutional settings. Gerontologist. 2001 Aug;41(4):462-73. doi: 10.1093/geront/41.4.462. PMID 11490044
- [Background] Girgis A, Sanson-Fisher RW, McCarthy WH. Communicating with patients: surgeons' perceptions of their skills and need for training. Aust N Z J Surg. 1997 Nov;67(11):775-80. doi: 10.1111/j.1445-2197.1997.tb04578.x. PMID 9396993
- [Background] Survey of Physician Attitudes Regarding the Care of Cancer Survivors (SPARCCS) [Internet]. [cited 2018 Feb 19]. Available from: https://healthcaredelivery.cancer.gov/sparccs/
- [Background] PASS 15 Power Analysis and Sample Size Software (2017). NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass.
- [Background] 95% Confidence Intervals for a Proportion [Internet]. Available from: http://web1.sph.emory.edu/cdckms/proportionDEFF.html
- [Background] Levy PS, Lemeshow S. Sampling of populations: methods and applications. 4th ed. Hoboken, N.J: Wiley; 2008. 576 p. (Wiley series in survey methodology).
- [Background] Lohr, Sharon. Sampling: Design and Analysis. Belmont, CA: Duxbury Press, 1999. Chapter 11.
- [Background] Applebaum AJ, Farran CJ, Marziliano AM, Pasternak AR, Breitbart W. Preliminary study of themes of meaning and psychosocial service use among informal cancer caregivers. Palliat Support Care. 2014 Apr;12(2):139-48. doi: 10.1017/S1478951513000084. Epub 2013 Aug 7. PMID 23919966
- [Background] Dionne-Odom JN, Applebaum AJ, Ornstein KA, Azuero A, Warren PP, Taylor RA, Rocque GB, Kvale EA, Demark-Wahnefried W, Pisu M, Partridge EE, Martin MY, Bakitas MA. Participation and interest in support services among family caregivers of older adults with cancer. Psychooncology. 2018 Mar;27(3):969-976. doi: 10.1002/pon.4603. Epub 2017 Dec 28. PMID 29226997
- [Background] Lund L, Ross L, Petersen MA, Groenvold M. The interaction between informal cancer caregivers and health care professionals: a survey of caregivers' experiences of problems and unmet needs. Support Care Cancer. 2015 Jun;23(6):1719-33. doi: 10.1007/s00520-014-2529-0. Epub 2014 Nov 29. PMID 25432867
- [Background] Mosher CE, Champion VL, Hanna N, Jalal SI, Fakiris AJ, Birdas TJ, Okereke IC, Kesler KA, Einhorn LH, Given BA, Monahan PO, Ostroff JS. Support service use and interest in support services among distressed family caregivers of lung cancer patients. Psychooncology. 2013 Jul;22(7):1549-56. doi: 10.1002/pon.3168. Epub 2012 Sep 3. PMID 22941782
- [Background] Condition-Specific Research | National Alliance for Caregiving [Internet]. [cited 2017 Oct 13]. Available from: http://www.caregiving.org/research/condition-specific/
- See also: [cited 2017 Oct 13] — http://www.caregiving.org/research/condition-specific/